CLINICAL TRIAL: NCT03926442
Title: Reason to Season: Flavors to Increase Vascular Health
Brief Title: Spices, Inflammation and Vascular Response in Humans
Acronym: SPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IRB2019-014
Record Dates: First submitted 2019-04-19; First posted 2019-04-24 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Healthy
Keywords: Spices; Herbs; Metabolic responses; Endothelial function; Inflammatory markers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active1 (Experimental): Italian Herb in active breakfast meal
  Interventions: Other: Italian Herb meal
- Active2 (Experimental): Cinnamon in active breakfast meal
  Interventions: Other: Cinnamon Meal
- Active3 (Experimental): Pumpkin Spice Mix in active breakfast meal
  Interventions: Other: Pumpkin Spice meal
- Placebo Comparator (Placebo Comparator): Placebo Breakfast
  Interventions: Other: Placebo meal

INTERVENTIONS:
Other: Italian Herb meal — Italian Herb in active breakfast meal
  Other Names: Italian Herb
  Arms: Active1
Other: Cinnamon Meal — Cinnamon in active breakfast meal
  Other Names: Cinnamon
  Arms: Active2
Other: Pumpkin Spice meal — Pumpkin Spice Mix in active breakfast meal
  Other Names: Pumpkin Spice Mix
  Arms: Active3
Other: Placebo meal — Placebo in breakfast meal
  Other Names: Placebo
  Arms: Placebo Comparator

SUMMARY:
The objectives of this study are:

1. To characterize the time course of herbs/spice action on endothelial function as measured by FMD over 24 h using a challenge meal paradigm.
2. To assess effects of herbs/spices on metabolic indices (ie., glucose, insulin), and inflammatory markers such as cytokines (ie., IL-6, TNF-alpha) and vascular adhesion molecules (ICAM and VCAM).

DETAILED DESCRIPTION:
The proposed study will be conducted in humans according to Good Clinical Practice (GCP) guidelines. All subjects will review and sign an Informed Consent Form approved by the Illinois Institute of Technology's Institutional Review Boards (IRB) prior to screening.

This single-center clinical trial is a randomized, blinded, 4-arm, placebo-controlled, within subject cross-over trial, featuring a repeated postprandial sampling paradigm to evaluate the effects of spice/herb intake on endothelial function, inflammation, insulin sensitivity / glucose handling and vascular function in overweight/obese adults after consuming a standardized challenge meal.

A planned sample size of 24 will be enrolled into the study. This study will require one initial screening visit and 4 study visits. This study will take approximately 4-5 weeks per subject to complete.

The initial screening visit will provide subject with their site-specific, IRB-approved informed consent document prior to the start of any study related procedures. Subject eligibility will be determined through anthropometric measurements, vital signs, fasting blood glucose test (finger prick), and completion of a survey relate to general eating, health, mood and exercise habits.

Eligible subjects will follow a limited polyphenolic diet throughout the duration of their participation, although stricter guidelines will be imposed during the 3 days prior to a study visit. Shopping lists and meal plans will be provided to subjects, along with counseling by our study dietitians, to help subjects adhere to the limited polyphenolic diet. The trial will initiate with a 3-day food diary to assess background (pre-study) dietary intake followed by counseling to follow a diet relatively low in (poly)phenolic rich-beverages/foods, which will be maintained for the duration of the experiment. After an initial 7-day run-in period on the limited polyphenolic diet, subjects will be randomized to 1 of 4 treatment sequences. Treatment codes will be maintained by the principal investigator/study physician. All subjects will receive four treatments, once each on 4 different occasions and separated by at least 4 days. Italian Herb mix, Cinnamon, Pumpkin Spice or placebo will be provided with a standardized meal.

Each visit will last ~8 hours and subjects will be required to remain at the Clinical Unit for the duration of the visit. Blood samples will be collected at 0 (fasting) and at 0.5 h, 1 h, 2 h, 4 h, 5.5 h, 7 h and 24 h via a catheter placed on the non-dominant arm by a registered nurse. FMD or NIRS will be conducted at the CNRC or the HNRCA, respectively at 0 (fasting) and at 1 h, 2 h, 4 h, 5.5 h, 7 h and 24 h.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 35 kg/m2
* Aged 18 years and older
* Able to provide informed consent and comply with study procedures
* Willing to maintain stable body weight and follow his/her habitual diet and physical activity patterns throughout the trial.
* Judged by the Investigator to be in general good health on the basis of medical history and screening laboratory tests.
* People with no documented disease condition that would interfere with the study endpoints (ie., CVD, diabetes, hypertension, major organ diseases) or taking medication or dietary supplements that may interfere with study endpoints

Exclusion Criteria:

* Current smoker or marijuana user
* No history or presence of atherosclerosis/cardiovascular disease, inflammatory disease, diabetes mellitus, or other systemic diseases, psychological or psychiatric disorders that may interfere with study outcomes.
* Taking any medications and/or supplements that would interfere with outcomes of the study (i.e., lipid-lowering medications, anti-inflammatory drugs, etc)
* Unstable use of any medication/supplement, this could include marijuana used as -needed for medical reasons
* Have a history of cancer, except for non-melanoma skin cancer in past 5 years
* Addicted to drugs and/or alcohol (>4 drinks/day)
* Have been exposed to any non-registered drug product within last 30 days.
* Working overnight (e.g. 3rd shift of overnight workers)
* Excessive exercisers or trained athletes
* Have allergies/intolerances to cinnamon, Italian herbs, etc.
* Extreme dietary habits (ie. vegetarian/vegan)
* Excessive coffee/tea drinker (>4 cups/day)
* Actively losing weight/ trying to lose weight (unstable body weight fluctuations of > 5 kg in 3 months)
* Donated blood within last 3 months
* Female who is pregnant, planning to be pregnant, breastfeeding
* Any condition the Investigator believes would interfere with his or her ability to provide informed consent or comply with the study protocol, or which might confound

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Changes in postprandial endothelial function among 4 treatments measured in percent flow mediated dilation | Baseline to 24 hours
  Vascular Assessments will be measured with Flow mediated vasodilation (FMD)

SECONDARY OUTCOMES:
Changes in Plasma Interleukin-1 β (IL-1β) concentration response among 4 treatments. | Baseline to 24 hours
  Inflammatory cytokines (Interleukin-1 β (IL-1β) will be measured using single target ELISA technology (R&D Systems).
Changes in Plasma Interleukin-6 (IL-6) concentration response among 4 treatments. | Baseline to 24 hours
  Inflammatory cytokines (Interleukin-6 (IL-6) will be measured using single target ELISA technology (R&D Systems).
Changes in Plasma Tumor Necrosis Factor-α (TNF-α) concentration response among 4 treatments. | Baseline to 24 hours
  Inflammatory cytokines (Tumor Necrosis Factor-α (TNF-α) will be measured using single target ELISA technology (R&D Systems).
Changes in Plasma intercellular adhesion molecule 1 (ICAM 1) concentration response among 4 treatments. | Baseline to 24 hours
  Inflammatory cytokines (intercellular adhesion molecule 1 (ICAM 1) will be measured using single target ELISA technology (R&D Systems).
Changes in Plasma vascular cell adhesion molecule 1 (VCAM 1) concentration response among 4 treatments. | baseline to 24 hours
  Inflammatory cytokines (vascular cell adhesion molecule 1 (VCAM 1)) will be measured using single target ELISA technology (R&D Systems).

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Huang Y, Edirisinghe I, Burton-Freeman BM, Sandhu AK. Characterization and Pharmacokinetic Profile of Herbs and Spices' Phytochemicals over 24 h after Consumption in Overweight/Obese Adults. Mol Nutr Food Res. 2023 Jul;67(14):e2200785. doi: 10.1002/mnfr.202200785. Epub 2023 Jun 13. PMID 37310415
- [Derived] Huang Y, Tsai MF, Thorat RS, Xiao D, Zhang X, Sandhu AK, Edirisinghe I, Burton-Freeman BM. Endothelial Function and Postprandial Glucose Control in Response to Test-Meals Containing Herbs and Spices in Adults With Overweight/Obesity. Front Nutr. 2022 Feb 22;9:811433. doi: 10.3389/fnut.2022.811433. eCollection 2022. PMID 35273988